CLINICAL TRIAL: NCT05334498
Title: Comparative Effects of Motor and Cognitive Dual-task Gait Training on Balance and Mobility in Persons With Intellectual Disabilities
Brief Title: Motor and Cognitive Dual-task Gait Training Effect Functional Outcome in Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah Maria Asghar /21923
Record Dates: First submitted 2022-02-20; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Intellectual Disability
Keywords: Motor and cognitive dual task gait training
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor dual-task gait training (Experimental): Motor dual task gait training was the protocol which performed by the patients after the measurement of the balance and gait ability
  Interventions: Other: Motor dual-task gait training
- Cognitive dual-task gait training (Experimental): Cognitive dual task gait training was the protocol which performed by the patients after the measurement of the balance and gait ability
  Interventions: Other: Cognitive dual-task gait training

INTERVENTIONS:
Other: Motor dual-task gait training — Patients were instructed to walk either on treadmill or on the land. During walk; patients were instructed to perform five tasks. The patients performed tossing and catching the ball, rehanging loops on hoops, buttoning and unbuttoning the shirts, holding the cup in water without the spilling and receiving with returning the water. Each activity were performed for three minute and 15 minutes were provided for performing all the tasks
  Arms: Motor dual-task gait training
Other: Cognitive dual-task gait training — Patients were instructed to walk either on treadmill or on the land. During walk; patients were instructed to perform five tasks. The patients performed sharp coloring, subtraction, counting, verbal analogical reasoning and backward spelling. Each activity were performed for three minute and 15 minutes were provided for performing all the tasks
  Arms: Cognitive dual-task gait training

SUMMARY:
To find out the comparative effects of motor and cognitive dual gait training on improving the balance control and mobility skills among intellectual disable patients.

DETAILED DESCRIPTION:
Previous studies had done a lot of work in improving balance and mobility skills by combining both motor and cognitive dual gait training (CDT and MDT) techniques among Down syndrome, Parkinsonism and so on but not a single study was conducted in order to determine the comparative effects of CDT and MDT especially in intellectual disability individuals to improve balance so the study was conducted in order to find the comparative effect for the better understanding of the treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Both genders having IQ range between 50-69
* Walk without assistive devices
* Having a Grade I-IV on the RLACFS

Exclusion Criteria:

* Genetic disorders (Down syndrome).
* Age-related diseases like Parkinsonism and Alzheimer disease.
* Cerebrovascular accident, dementia, Cerebral palsy
* Severe visual impairment.
* Medications (sedatives or narcotics)

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Rancho Los Amigos Cognitive functional scales | 4th week
  Ranchos Los Amigos Scale is the reliable tool for assessing the cognitive function of the patient as the scale score form grade 1 to 8 with ten level descriptive scale where grade 1 have zero response while grade 8 shows the activate participation of the patient with cut off value for 5. It is the most reliable and valid assessment tool
Berg Balance Scale | 4th week
  Berg Balance Scale is the most reliable tool used for the assessment of balance performance among patients having balance problems and disease causing balance issues.
Walking while talking test | 4th week
  Walking while talking is the time measuring tool for assessing the risk of fall and gait performance in the intellectual disable patients as in this test the patient asked to narrate repeated words during walking for 20 feet having ICC= 0.89-0.99
Stair climb test | 4th week
  Stair climbing test is the valid tool for assessing the velocity and level of mobility within the time as the patient asked to climb up and down the stairs and therapist record the number of the steps which are taken within the time period having MIC of -0.6 with 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, MSPT, Principal Investigator — Riphah International University
Locations (1):
- District headquarter hospital, Mirpur, Azad Jammu Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No